CLINICAL TRIAL: NCT00967915
Title: Efficacy of Neonatal Release of Ankyloglossia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007.0077
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Ankyloglossia
Keywords: Ankyloglossia; Tongue tie; Frenotomy; Frenulectomy; Breast feeding; HATLFF; IBFAT
MeSH Terms: conditions — Ankyloglossia; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Frenotomy (Experimental): Group of neonates that will receive frenotomy for tongue-tie
  Interventions: Procedure: Frentomy
- No frenotomy (Sham Comparator): Group of infants that will undergo sham procedure (no frenotomy performed)
  Interventions: Other: Sham procedure

INTERVENTIONS:
Procedure: Frentomy — Frenotomy will be performed. This procedure involves crushing frenulum tissue with straight hemostat for hemostasis and anesthesia while tongue is elevated with elevator. Frenulum then cut to desired length with iris scissors. Patient then returned to parents and immediately breastfeeds without parent observing infant's mouth.
  Arms: Frenotomy
Other: Sham procedure — Infant taken into room away from parents and no frenotomy performed. Infant's mouth is examined but no interventions made.
  Arms: No frenotomy

SUMMARY:
The purpose of this study is to determine if frenotomy for ankyloglossia will improve infant breastfeeding, decrease maternal nipple pain and increase duration of breastfeeding with the hypothesis that frenotomy will do all of the above.

DETAILED DESCRIPTION:
The primary objective of our study is to determine if frenotomy (or release of tongue tie) for ankyloglossia (tongue tie) will decrease maternal nipple pain with breast feeding and improve infant's ability to breast feed. Our secondary objective is to determine if frenotomy for ankyloglossia will improve the length of time a mother breast feeds. Our hypothesis is that frenotomy will decrease maternal nipple pain, improve infant's breast feeding and prolong the duration of breast feeding.

ELIGIBILITY:
Inclusion Criteria:

* Significant ankyloglossia as judged by Hazelbaker scale (HATLFF)
* Report of maternal nipple pain with feeding
* Report of difficulty with infant breast feeding

Exclusion Criteria:

* Significant craniofacial defects
* Age >14 days at enrollment
* Any maternal contraindication to breastfeeding
* Neurologic defects that would impair breast feeding

Ages: 0 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2007-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Maternal nipple pain as judged by R. Melzack's short form pain scale and infant breast feeding as judged by IBFAT scale | immediately following 1st breast feed, and at 2 week, 2,4,6 12 month follow ups

SECONDARY OUTCOMES:
Length of breast feeding | 1 year follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center Portsmouth, Portsmouth, Virginia, United States

REFERENCES:
- [Derived] Buryk M, Bloom D, Shope T. Efficacy of neonatal release of ankyloglossia: a randomized trial. Pediatrics. 2011 Aug;128(2):280-8. doi: 10.1542/peds.2011-0077. Epub 2011 Jul 18. PMID 21768318